CLINICAL TRIAL: NCT02510638
Title: The Clinical Epidemiology of Hospitalized Dengue Cases in Malaysia
Status: Completed | Type: Observational
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Woon Yuan Liang, Doctor, Clinical Research Centre, Malaysia
Other Study IDs: NMRR-15-452-25624
Record Dates: First submitted 2015-07-26; First posted 2015-07-29 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dengue infection has been identified as the fastest spreading mosquito-borne viral disease by World Health Organization (WHO), which affects more than 2.5 billion people living in the subtropical and tropical regions. Malaysia is hyper-endemic with all four dengue virus serotypes circulating and responsible for the escalating number of cases over the years. As of 28 February 2015, there are 62 deaths secondary to dengue infection being reported in Malaysia; and the total number of dengue cases reported in the same period was 23,966 which is 46% higher than the same reporting period of 2014. Although dengue virus has been identified for so many years and plenty of research work has been carried out, it was proven that there are still many aspects that we are not too sure about the disease. Therefore, this multi-center, observational cohort study is designed to investigate the clinical course of hospitalized dengue infection in Malaysia. The study population of this study consists of male or female patients with dengue to be randomly sampled from hospitals in Malaysia. This study will be conducted in 2 stages whereby the 1st stage will only focus on the basic social and clinical data to describe the clinical course of dengue as general and the 2nd stage will collect the more detailed clinical and management data to describe the detailed clinical course, management and prognosis of dengue. All hospital participation in this study is voluntary, and approval will be obtained from National Institute of Health (NIH) and Medical Research Ethics Committee (MREC) prior to any recruitment.

DETAILED DESCRIPTION:
Dengue infection have resurged and disseminated globally since late 1970s after successful eradication programs of the dengue vector Aedes mosquitoes in Latin America in the 1940s. It has been identified as the fastest spreading mosquito-borne viral disease by World Health Organization (WHO), which affects more than 2.5 billion people living in the subtropical and tropical regions. Approximately 75% of the current global dengue disease burden comes from the population residing at Southeast Asia and Western Pacific regions, which subsequently lead to the formation of the Asia Pacific Dengue Strategic Plan (2008-2015) and the recent Global Strategy for Prevention and Control (2012-2020) to reduce the dengue burden.

Malaysia is hyper-endemic with all four dengue virus serotypes circulating and responsible for the escalating number of cases over the years. The number of reported dengue cases in Malaysia has increased fourfold from 44.3 per 100,000 population in 1999 to 181 per 100,000 in 2007; with increased in dengue deaths in the adult populations since 2002. Worst still, as of 28 February 2015, there are 62 deaths secondary to dengue infection being reported in Malaysia; and the total number of dengue cases reported in the same period was 23,966 which is 46% higher than the same reporting period of 2014.

The WHO has revised the dengue classification in 2009, which were shown to be more sensitive than the WHO 1997 classification system in predicting severity of dengue. According to this WHO 2009 classification, dengue infection is now categorized into dengue, dengue with warning signs, and severe dengue. The proposed warning signs include abdominal pain or tenderness, persistent vomiting, clinical fluid accumulation, mucosal bleed, lethargy or restlessness, liver enlargement > 2cm, increase in hematocrit concurrent with rapid decrease in platelet count. Severe dengue is then defined as dengue infection with severe plasma leakage with shock, severe bleeding or severe organ involvement.

Although a large number of patients may recover from this self-limiting disease, a small proportion may progress to develop severe dengue manifestations, which requires admission to intensive care unit (ICU) for closer monitoring and intervention. However, the progression to severe clinical manifestations is usually unpredictable. Early identification of signs that can predict severe dengue may save lives by facilitating early initiation of interventions and frequent monitoring. Dengue epidemics in Malaysia lead to a strong demand for hospital beds and manpower, and inflicting large public and private hospitalization costs. Hence, it is crucial to determine a predictive tools which can help to triage patients into those that are least and most likely to develop complications in order for a better allocation of limited healthcare resources.

A few studies have been done to validate the utility of the proposed warning signs by WHO 2009 dengue classification, but the results vary and none of these studies are conducted in our local setting. Although dengue virus has been identified for so many years and plenty of research work has been carried out, it was proven that there are still many aspects that we are not too sure about the disease. It got more confused with the sudden surge of dengue cases and dengue mortality cases since last year. Therefore, this study aims to look into the clinical course of the hospitalized dengue cases in Malaysia. It will then allow us to zoom in to the specific area for more future research work.

General Objective:

To study the clinical course of hospitalized dengue cases in Malaysia in from year 2009 till 2015.

Specific Objectives are to:

1. Describe the characteristics of patients hospitalized for dengue
2. Describe the clinical presentation of patients hospitalized for dengue
3. Verify the diagnosis of reported dengue cases
4. Describe the spectrum of disease severity among patients hospitalized for dengue
5. Describe the management of patients hospitalized for dengue including ICU care
6. Describe the prognosis of patients hospitalized for dengue
7. Estimate the resource utilization and cost of care of patients hospitalized for dengue
8. Estimate the mortality outcome of patients hospitalized for dengue

This will be a multi-center, observational cohort study designed to investigate the clinical course of patients hospitalized for dengue infection in Malaysia. This study will be conducted in 2 stages for the duration of 6 months. Data will be retrieved retrospectively in both stages.

In Stage 1, a sample of dengue cases who visited general practitioner or who were hospitalized in from year 2009 until 2015 will be sampled using PIK and Health insurance claims database as sampling frame. Each hospital will be given a list of the dengue cases and the local coordinator from respective hospital Clinical Research Centre (CRC) will trace the medical records of all these dengue cases. Once the case notes of all the dengue cases are traced, two trained research assistants will travel to the hospital to extract the basic clinical data on social demographics, presentation and discharge status by using case report form A. All the data collected in phase 1 will be categorized as basic clinical set.

In Stage 2, a subset of the basic clinical set will be sampled conveniently. Only the cases that were tested positive by dengue non-structural protein 1 (NS1), immunoglobulin-M (IgM) or high-titre immunoglobulin-G (IgG) will be included in the Stage 2 study. A more detailed clinical subset data will be collected by research assistants at site. All co-morbidity, serial clinical and laboratory data, in-hospital course and treatment data and Intensive Care Unit (ICU) admission data will be extracted from medical records with case report form B. All variables/data in the case report form is defined in Appendix I. All data collected in Stage 1 and 2 will then be compiled and analyzed with software Stata Version 10.0.

WHO 2009 classification will be adopted in this study. According to the WHO 2009 criteria, probable dengue is defined as fever and two of the following: nausea or vomiting, rash, aches and pain, leucopenia, and any warning signs. Warning signs are abdominal pain or tenderness, persistent vomiting, clinical fluid accumulation, mucosal bleed, lethargy or restlessness, hepatomegaly and hematocrit changes ≥20% concurrent with platelet <50,000 on the same day. Severe dengue is present if any of the following criteria fulfilled:

I) Plasma leakage evidenced by hematocrit change of ≥20%, pleural effusion or ascites, or hypoproteinemia, leading to:

* Dengue shock syndrome (tachycardia, cold and clammy extremities, capillary refill time greater than 3 seconds, weak or undetectable pulse, narrow pulse pressure ≤20 mmHg, or systolic blood pressure <90 millimetre mercury (mmHg) or unrecordable blood pressure); or
* Fluid accumulation with respiratory distress (respiratory rate ≥30/minute, oxygen saturation ≤92% on room air, or mechanical ventilation) II) Severe bleeding manifesting as gastrointestinal bleeding or menorrhagia, or requirement for transfusion of packed red blood cells or whole blood.

III) Severe organ involvement as follows:

* Serum alanine or aspartate transaminase ≥1000 units/L;
* Impaired consciousness;
* Acute renal impairment defined as serum creatinine > two times upper limit of normal;
* Myocarditis or encephalopathy/encephalitis

ELIGIBILITY:
Inclusion Criteria:

* Stage 1:

  * Discharge diagnosis with International Classification of Disease (ICD) code A90 - A99
  * Availability of minimal dataset (name, IC, age, sex, diagnosis, date admit, date discharge, discharge status)
* Stage 2:

  * Laboratory confirmed dengue (Non-structural 1 antigen, dengue IgM, high-titre dengue IgG, and dengue polymerase chain reaction (PCR) positive)

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of male or female patients with Dengue to be randomly sampled from hospitals in Malaysia. Approximately 384 patients will be enrolled.
  Sampling Frame: A sample of dengue cases who visited general practitioner or who were hospitalized from year 2009 till 2015 will be sampled using PIK and Health insurance claims database. Sampling: A random sampling will be done to select the samples. In order to do it, each subject in the sampling frame will be given an unique number (e.g.: 001, 002, 003,… etc) according to the sequence of notification date. Then, the subjects will be selected randomly by using randomizer.org software.
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with severity of disease | Participants will be observed for the period of hospital stay, for an average of 1 week duration

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Hospital Kuala Lumpur, KualaLumpur, Malaysia